CLINICAL TRIAL: NCT02734511
Title: Efficiency and Safety of a Procedural Sedation by Propofol Administered by Trained Doctors Who Are Not Anesthesiologists on Terminally Ill Patients With Refractory Pain Hospitalized in a Palliative Care Unit
Brief Title: Efficiency and Safety of a Procedural Sedation by Propofol on Terminally Ill Patients With Refractory Pain
Acronym: PROPOPAL2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-AOI-07
Record Dates: First submitted 2016-03-31; First posted 2016-04-12 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2023-11

CONDITIONS: Refractory Pains
MeSH Terms: conditions — Pain, Intractable | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug: sedation with propofol (Experimental): induction with propofol at 20mg/kg/h. Then, when the patient is sleeping, dosage is decreased to 6 mg/kg/h
  Interventions: Drug: sedation with propofol

INTERVENTIONS:
Drug: sedation with propofol — induction with propofol at 20mg/kg/h. Then, when the patient is sleeping, dosage is decreased to 6 mg/kg/h

SUMMARY:
Relieving symptoms of patients hospitalized in a palliative care unit is a priority. Although they receive appropriate care, they may still experience pain refractory to analgesia or/and to conservative treatment during care procedures. For instance, pain can be caused by the bandaging of carcinological or ischemic wounds, or by the mobilization of traumatic injuries which cannot be specifically treated.

Although these types of situations are rare, they remain unacceptable, especially at the end of life.

According to current recommendations, a short-term sedation treatment can be administered although detailed procedures for this type of sedation have not been very much documented. In reality, midalozam is often used in those cases but it has drawbacks, which is why the investigators have looked into alternatives.

Propofol, which is already widely used in anesthesia and emergency medicine to manage painful procedures, seems to be an interesting molecule because of its pharmacological properties. It allows to quickly reach deep sedation and thus obtain a certain level of comfort for the patient, but also ensures a prompt awakening as soon as care procedures are over, which limits respiratory side effects.

The results from a preliminary study encouraged us to go further and to present a prospective study conducted in multiple centers in order to evaluate the efficiency and safety of a procedural sedation administered by trained doctors who are not anesthesiologists on terminally ill patients with refractory pain hospitalized in a palliative care unit.

DETAILED DESCRIPTION:
At the end of life, some patients may feel pain during care procedures. These painful procedures contribute to the patient's overall suffering. Of course the investigators do not take into account procedures which could be considered as futile medical care and would not bring any comfort to the patient. The procedures that the investigators do consider are necessary and acceptable: basic hygiene care, such as bandaging. Even with the best palliative care, certain pains caused by these procedures can be refractory to analgesics, to Entonox and to other conservative treatments. These pains are ethically unacceptable, especially at the end of life. In these cases, short-term procedural sedation could benefit the patient, as indicated by the Agence Nationale de Sécurité du Médicament (French Agency for the Safety of Health Products). However, there are no documented recommendations on the way to administer these types of sedations because of a lack of scientific studies in that field. It therefore remains an important issue in palliative care research. The sedations consist of a transitory reduction of vigilance which is sufficient enough for the patient not to suffer. They are therefore a major tool to provide sufficient comfort to terminally ill patients while being used as part of a treatment approach. However, they still have drawbacks: patients lose contact with the environment but can also experience respiratory complications (embarrassment, respiratory depression, inhalation). These risks compel the investigators to only use these sedations for terminally ill patients suffering from major refractory pain at the end of life, in which case they consider that comfort is an absolute priority (principle of double effect). The decision to use sedation must be agreed upon after collegial consultation and discussion with the patient and/or his or her relatives. The risk of side effects must be reduced as far as possible without pursuing a reanimation approach which would go against a palliative approach.

Sedation, which was originally exclusively administered by anesthesiologists, has been used by palliative care doctors for many years. At first, midazolam seemed to be the best sedative agent and its use spread although it has not been much documented in that context. However, midazolam has its limits. It cannot provide a very deep sedation because of its respiratory depressant effect and the patient, when under light sedation, often experiences persistent discomfort. Moreover, midazolam requires a long titration period and often causes a sedation which can last several hours, thus reducing the patient's relational life and increasing the risk of congestion and respiratory depression. Investigators are therefore looking for alternatives. According to them, propofol would be a suitable molecule because of its pharmacological properties. Its pharmacokinetic properties allow the patient not only to quickly reach deep sedation and therefore better comfort, but also to wake up as soon as the painful care procedure is completed, thus limiting the risk of respiratory side effects.

Note that it is already used in other situations for procedural sedation by doctors who are not anesthesiologists (pulmonologists, gastroenterologists, emergency doctors).

In a feasibility study, investigators pointed out that propofol could be used in a palliative care unit for transitory sedation administered by an anesthesiologist following a strict protocol and could relieve terminally ill patients at the end of life during painful care procedures in a sufficiently safe way (preliminary results presented at the French Society of Support and Palliative Care conference in 2015).

Investigators aim at showing that a procedural sedation using propofol can be administered by palliative care doctors who are not anesthesiologists but have been trained to follow a precise protocol and that it can bring relief to terminally ill patients with refractory pain experienced during care procedures without causing major side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in the palliative care unit
* Patient whose prognosis is three months or less life expectancy
* Patient treated with step 3 opioids
* Pain experienced during care procedures and refractory to transmucosal fentanyl and equimolar mixture of oxygen and nitrous oxide if the latter is not contraindicated
* The pain scales used are Numeric Rating Scale ≥ 3/10 for patients able to communicate and Algoplus scale > 2 for patients with inability to communicate verbally
* Indication of procedural sedation is agreed upon after collegial consultation and evaluation of the benefit risk balance (principle of double effect)
* Age: 18 and above
* Patient must be registered for social security
* Consent must be signed before and by the conscious patient or by his or her trusted person or relative for patients with cognitive impairments or disturbed vigilance

Exclusion Criteria:

* contra-indication to soya
* contra-indication to egg lecithin
* Respiratory insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
success rate of care without severe pain for the patient | from the beginning of sedation to 2 hours after sedation
  Success is defined as the administration of care without severe pain for the patient
success rate of care without major side effects | from the beginning of sedation to 2 hours after sedation
  Major side effects are defined as ''Sentinel AEs'' by the World SIVA (Society of IntraVeinous Anesthesia) International Sedation Task Force

CONTACTS AND LOCATIONS:
Overall Officials: Flora TREMELLAT, MD, Principal Investigator — Unité de Soins Palliatifs, CHU de Nice
Locations (1):
- CHU de Nice - Hôpital de l'Archet, Nice, Alpes-Maritimes, France

IPD SHARING:
Plan to Share IPD: No